CLINICAL TRIAL: NCT02438839
Title: Curative Chemoradiation of Low Rectal Cancer. A Prospective Multicenter Observational Study
Brief Title: Curative Chemoradiation of Low Rectal Cancer
Acronym: WW2
Status: Active, not recruiting | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WW2
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the present study is to investigate whether curative chemoradiation of low rectal cancer is feasible, safe and effective in a multicenter study with results comparable to those of single center studies.

Results from previous studies indicate that a considerable fraction of patients with low rectal cancer can be cured by a combination of radiation and chemotherapy alone and thus be spared from operation.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified adenocarcinoma of the rectum
* Planned abdominoperineal resection (APR) or ultralow resection
* Primary, resectable T1-T3, N0 tumor. N1 nodal disease is acceptable, if the positive lymph nodes are localized to the mesorectum at the level of the tumor.
* Distance from anal verge to lower edge of tumor ≤ 6 cm measured by rigid rectoscope
* Performance status 0-2
* Patient acceptance to collection of biopsies and blood samples for translational research
* Age ≥ 18 years
* Normal function of bone marrow as evaluated by

  * neutrophils ≥ 1.5 x 10^9/l
  * thrombocytes ≥ 100
* Normal function of liver

  * alanine aminotransferase (ALAT) < 2.5 x upper limit of normal
  * bilirubin < 2.5 x upper limit of normal
* Kidney function

  - Serum creatinine < 1.5 x upper limit of normal or measured glomerular filtration rate (GFR) > 30 ml/min
* Fertile women must present a negative pregnancy test and use secure contraceptives during and 3 months after treatment.
* Written and orally informed consent

Exclusion Criteria:

* Previous surgical treatment of the present cancer, including transanal excision of tumor.
* Other malignant disease within the past five years except basocellular skin cancer and carcinoma in situ cervicis uteri
* Distant metastases verified by imaging or biopsy
* Previous radiation treatment of the pelvis
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low rectal cancer (tumor located ≤ 6 cm from the anal verge) who are referred to the participating departments and who fulfill the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with locoregional tumor control with chemoradiation alone two years after end of treatment | 2 years after end of treatment

SECONDARY OUTCOMES:
Cumulative incidence of local recurrence after surgery | Every two months the first year, every three months the second year, every six months the third year, and annually the fourth and fifth years
Rate of distant metastases | Every two months the first year, every three months the second year, every six months the third year, and annually the fourth and fifth years
Response and tumor control on MRI scans compared to clinical observations, including rectoscopic examination | 6 and potentially 12 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Department of Oncology, Vejle Hospital; Henrik Jensen, PhD, Principal Investigator — Department of Oncology, Vejle Hospital
Locations (5):
- Denmark (5):
  - Department of Oncology, Aalborg University Hospital, Aalborg
  - Department of Surgery, Aalborg University Hospital, Aalborg
  - Department of Oncology, Rigshospitalet, Copenhagen
  - Department of Oncology, Vejle Hospital, Vejle
  - Department of Surgery, Vejle Hospital, Vejle